CLINICAL TRIAL: NCT01781442
Title: An Open Label, Non-interventional Study Of The Safety Of Temsirolimus Injection (Torisel) In The Treatment Of Advanced Renal Cell Carcinoma In Filipino Adult Patients: A Post Marketing Surveillance Study
Brief Title: A Post Marketing Surveillance As Required By Philippine Food And Drug Administration
Status: Withdrawn | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1771110
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — temsirolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient Arm- temsirolimus
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — The recommended dose of Torisel is 25 mg infused over a 30-60 minute period once a week.
  Treatment will continue until disease progression or unacceptable toxicity.
  The use and dosage recommendations for Torisel will take place on the basis of the approved local product document and will be adjusted solely according to medical and therapeutic necessity.

SUMMARY:
This is a post marketing surveillance which determines the safety profile of the product to Filipinos. This is a FDA requirement for registration.

DETAILED DESCRIPTION:
The Philippine Food and Drug Administration requires that a post marketing surveillance study be conducted nationwide and enroll approximately 3,000 study patients. In cases where the 3,000 patients will not be met, the total sample size can be reduced to 10% of the volume of drug use during the first year of it being marketed. Final sample size will be determined after one year of marketing authorization. The decision to use Torisel must be a joint decision made by the subject and the investigator.

The investigator must discuss product information with the subject as per usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that will be included in this post marketing surveillance study must be consistent with the approved label indication of Torisel in the Philippines.
* As per approved label indication, patients diagnosed with advanced renal cell carcinoma will be the ones eligible to participate in the study.
* The decision to prescribe Torisel will necessarily precede and will be independent of the decision to enroll the patient into the study.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Subjects with conditions that are contraindicated with Torisel based on the approved local product document in the Philippines will be excluded in this study. This condition includes: Patients with bilirubin >1.5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational, non-interventional study which will evaluate Torisel in Filipino adult subjects. Because the data to be collected will be under routine clinical conditions, subjects who have any of the contraindications specified in the product package insert are to be excluded. Torisel will be prescribed and administered according to the approved product information of the drug in the Philippines. Pfizer will not provide the drug for this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events [AEs] and Serious Adverse Events [SAEs] | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1771110&StudyName=A%20Post%20Marketing%20Surveillance%20As%20Required%20By%20Philippine%20Food%20And%20Drug%20Administration